CLINICAL TRIAL: NCT06948578
Title: Effectiveness and Safety of Thread-Embedding Acupuncture in Improving Functional Capacity and Quality of Life in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Thread-Embedding Acupuncture for Functional and QoL Improvement in COPD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Natasha Setiawan, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 25-04-0473
Record Dates: First submitted 2025-04-22; First posted 2025-04-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Chronic Pulmonary Obstruction
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: The intervention group will receive TEA, while the control group will receive sham TEA.
Who Masked: Participant, Outcomes Assessor
Masking Description: Blinding will be applied to participants and outcome assessors. Group allocation will not be disclosed to them to minimize assessment bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Thread-embedding acupuncture
  Interventions: Device: Thread embedding-acupuncture
- Control group (Sham Comparator): Sham thread-embedding acupuncture
  Interventions: Device: Sham thread-embedding acupuncture

INTERVENTIONS:
Device: Thread embedding-acupuncture — TEA is performed once at bilateral ST36 (perpendicular insertion) and BL13 (oblique insertion toward EX-B1) using absorbable PDO thread (CARA® 30G × 38 mm). Standard aseptic procedures are followed. Bleeding is controlled, and insertion sites are covered. Participants continue their routine pharmacological COPD treatment.
  Arms: Intervention Group
Device: Sham thread-embedding acupuncture — Sham TEA involves taping needles onto the surface of bilateral ST36 and BL13 without skin penetration or thread insertion. The direction toward EX-B1 is mimicked without actual insertion. All procedures, including marking and aseptic preparation, are performed identically to maintain blinding. Participants continue their routine pharmacological COPD treatment.
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to learn if thread-embedding acupuncture (TEA) can improve functional capacity and quality of life of chronic pulmonary disease (COPD) patients. The main questions it aims to answer are:

* Does TEA, when combined with standard treatment, improve functional capacity measured by the six-minute walking test (6MWT) and the modified Medical Research Council (mMRC) scale at 1, 2, and 3 months after the intervention?
* Does TEA, when combined with standard treatment, improve quality of life as measured by the COPD Assessment Test (CAT) and the St. George's Respiratory Questionnaire (SGRQ) at 1, 2, and 3 months after intervention? Researchers will compare TEA to sham TEA (a placebo procedure without thread implantation) to determine if TEA leads to meaningful improvements in COPD patients.

Participants will:

* Complete assessment using 6MWT, mMRC, CAT, and SGRQ
* Receive one session of either TEA or sham TEA
* Return to the clinic once a month for follow-up assessments over a 3-month period

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants aged 18 to 70 years.
* Body Mass Index (BMI) ≥18.5 kg/m².
* Diagnosed with stable chronic obstructive pulmonary disease (COPD) based on GOLD criteria.
* Willing to participate in the study until completion and has signed informed consent.

Exclusion Criteria:

* Pregnant women.
* Presence of tumors, wounds, inflammation, or skin infection at the needling area.
* Blood disorders or use of blood-thinning medications (antiplatelets or anticoagulants) with INR > 2.0.
* Uncontrolled heart disease or diabetes.
* Capillary blood glucose level ≥200 mg/dL (measured using glucometer).
* History of malignancy, uncontrolled epilepsy, or psychiatric disorders.
* Known allergy to stainless steel or polydioxanone (PDO) thread.
* Undergoing acupuncture therapy within the last 2 weeks or thread-embedding acupuncture (TEA) within the last 6 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Six-minute walking test (6MWT) | Baseline, 1 month, 2 months, 3 months after intervention
  Functional capacity will be assessed using the six-minute walking test (6MWT), measured as the distance (in meters) walked in six minutes.
Modified Medical Research Council (mMRC) Dyspnea Scale | Baseline, 1 month, 2 months, 3 months after intervention
  Dyspnea will be evaluated using the mMRC scale, scored from 0 to 4 based on the degree of breathlessness.
COPD Assessment Test (CAT) Score | Baseline, 1 month, 2 months, 3 months after intervention
  Health status and quality of life will be assessed using the CAT questionnaire, scored from 0 to 40.
  Higher scores indicate worse health status.
St. George's Respiratory Questionnaire (SGRQ) Score | Baseline, 1 month, 2 months, 3 months
  Quality of life will be evaluated using the SGRQ, which includes symptoms, activity, and impact domains.
  Scores range from 0 to 100, with higher scores indicating poorer quality of life.

SECONDARY OUTCOMES:
Frequency of Acute Exacerbation | From baseline to 3 months post-intervention
  The number of acute exacerbation events of COPD will be recorded over the study period.
Time to First Acute Exacerbation | From baseline to 3 months post-intervention
  Time (in days) from intervention to the first recorded acute exacerbation of COPD will be measured.
Frequency of Hospitalization | From baseline to 3 months
  The total number of hospital admissions due to COPD-related causes will be documented.
Duration of Hospitalization | From baseline to 3 months
  The cumulative duration (in days) of hospitalization related to COPD will be recorded.
Adverse Events Related to Intervention | Immediately post-intervention until 3 months
  Any adverse events occurring after the intervention, including infection, pain, or skin irritation at the insertion site, will be monitored and recorded.

CONTACTS AND LOCATIONS:
Overall Officials: KPEK FKUI-RSCM, Principal Investigator — The Health Research Ethics Commitee - Faculty of Medicine Universitas Indonesia and Dr. Cipto Mangunkusumo National Hospital
Locations (1):
- Universitas Indonesia, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No